CLINICAL TRIAL: NCT00728221
Title: Evaluation and Standardization of Ginseng and it's Components for Blood Pressure Regulation
Acronym: ESGC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 118328
Record Dates: First submitted 2008-08-01; First posted 2008-08-05 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Blood Pressure; Endothelial Function
Keywords: Ginseng; Korean Red Ginseng; Ginsenoside; Flow Mediated Dilation; Endothelial Function; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Asian ginseng; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo capsules (3g)
  Interventions: Dietary Supplement: Cornstarch
- 2 (Experimental): Whole Korean Red Ginseng root (3g)
  Interventions: Dietary Supplement: Korean Red Ginseng
- 3 (Experimental): Ginsenoside fraction of Korean Red Ginseng B (0.22g); bioequivalent to the original whole KRG root
  Interventions: Dietary Supplement: Korean Red Ginseng (Panax ginseng)
- 4 (Experimental): Polysaccharide fraction of KRG root (0.21g); bioequivalent to the original whole KRG root
  Interventions: Dietary Supplement: Korean Red Ginseng (Panax Ginseng)

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng — Cultivated KRG-B (central body Korean Red Ginseng) obtained from Kyonggi-do Farm, Kyonggi-do Province, Korea.
  Dosage form: whole root in capsules (3g)
  Other Names: Kyonggi-do Farm; C. A. Meyer
  Arms: 2
Dietary Supplement: Korean Red Ginseng (Panax ginseng) — Cultivated KRG-B (central body Korean Red Ginseng) obtained from Kyonggi-do Farm, Kyonggi-do Province, Korea.
  Dosage form: total ginsenoside fraction in capsules
  Other Names: Kyonggi-do Farm; C. A. Meyer
  Arms: 3
Dietary Supplement: Cornstarch — Placebo
  Arms: 1
Dietary Supplement: Korean Red Ginseng (Panax Ginseng) — Cultivated KRG-B (central body Korean Red Ginseng) obtained from Kyonggi-do Farm, Kyonggi-do Province, Korea.
  Dosage form: total polysaccharide fraction (panaxans) in capsules
  Other Names: Kyonggi-do Farm; C. A. Meyer
  Arms: 4

SUMMARY:
Ginseng has been used for many years in a wide array of anecdotal medicinal properties. Animal and limited clinical research points to the vascular effects of Korean Red Ginseng (KRG). The present project aims to assess the efficacy of KRG and contribution of its factionated components on various indices of vascular function in healthy individuals. Our primary objective is to compare the acute effects of KRG and placebo on endothelial function. Moreover, our secondary objective is to evaluate the effect of isolated KRG factions on arterial stiffness, blood pressure and vasoactive markers. We hypothesize that (1) consumption of KRG will cause an improvement in endothelial function in healthy individuals, as compared to placebo; (2) consumption of KRG will cause an improvement in arterial stiffness and blood pressure in healthy individuals, as compared to placebo; (3) the ginsenoside faction of KRG is primarily responsible for the anticipated vascular effects.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 70 years of age
* Healthy individuals (absence of major illnesses)

Exclusion Criteria:

* Primary hypertension (defined by the use of antihypertensive agents or a seated systolic blood pressure greater than or equal to 140mmHg or diastolic blood pressure greater than 90mmHg)
* Secondary hypertension (defined as SBP greater than 180mmHg and DBP greater than 110mmHg)
* Grade 3 hypertension (defined as SBP greater than 180mmHg and DBP greater than 110mmHg)
* Diabetes
* Chronic kidney disease
* Liver disease
* Estrogen-sensitive cancer
* Heavy alcohol use
* Bleeding disorders
* Planned surgery
* Angina
* CHF
* Coronary revascularization
* Peripheral vascular disease
* Coronary/cerebrovascular event in the last 6 months
* Prescriptions of MAO inhibitors, SSRIs, diuretics, sympathomimetics, herbal therapies, medication affecting nitric oxide synthesis, and/or anticoagulent medications within the last 6 months
* Sensitivity to any of the ingredients in the treatments or placebo
* Chronic use of or frequent prescriptions for NSAIDs
* Women of childbearing potential must not be pregnant or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the brachial artery | Start and finish of each treatment arm

SECONDARY OUTCOMES:
Augmentation Index | Start and finish of each treatment arm
Nitric Oxide and Cyclic GMP | Beginning of and 3 hours into clinical visit

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — St. Michael's Hospital, University of Toronto; Alexandra Jenkins, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Jovanovski E, Peeva V, Sievenpiper JL, Jenkins AL, Desouza L, Rahelic D, Sung MK, Vuksan V. Modulation of endothelial function by Korean red ginseng (Panax ginseng C.A. Meyer) and its components in healthy individuals: a randomized controlled trial. Cardiovasc Ther. 2014 Aug;32(4):163-9. doi: 10.1111/1755-5922.12077. PMID 24758417
- [Result] Jovanovski E, Jenkins A, Dias AG, Peeva V, Sievenpiper J, Arnason JT, Rahelic D, Josse RG, Vuksan V. Effects of Korean red ginseng (Panax ginseng C.A. Mayer) and its isolated ginsenosides and polysaccharides on arterial stiffness in healthy individuals. Am J Hypertens. 2010 May;23(5):469-72. doi: 10.1038/ajh.2010.5. Epub 2010 Feb 4. PMID 20134405